CLINICAL TRIAL: NCT01598181
Title: Transcranial Direct Current Stimulation (tDCS) as Treatment Method for Pain in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/2256/REK n; UNorthNorway (Other Grant/Funding Number: UNorthNorway)
Record Dates: First submitted 2012-03-15; First posted 2012-05-15 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2016-06

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active tDCS (Experimental)
  Interventions: Device: tDCS NeuroConn DC-stimulator plus
- sham tDCS (Sham Comparator): tDCS fades out after 20 sec. administered double blind by coded program.
  Interventions: Device: tDCS NeuroConn DC-stimulator plus; Device: sham tDCS

INTERVENTIONS:
Device: tDCS NeuroConn DC-stimulator plus — Anodal tDCS, M1, cathode supraorbital left, 2 mA, 20 min, 5 consecutive days.
  Other Names: model 0021; serial-no 0337
Device: sham tDCS — similar montage and time as active. Stimulation fades out after 20 sec.
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to investigate Transcranial Direct Current Stimulation as treatment method for pain in fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FIM) is a chronic pain condition with high prevalence. Studies involving neuroimaging techniques have identified functional differences in cerebral pain processing in patients with FIM, as compared to healthy controls. This may support that FIM do have a functional CNS component.

Transcranial Direct Current Stimulation (tDCS) is a non-invasive and safe method for inducing changes in cortical excitability. Previous studies showed that anodal stimulation of M1 may change pain perception, possibly by modulating functional anomalies in the FIM brain. The present study has two main goals:

1. To investigate if tDCS may provide FIM patients with symptom relief due to reduction of pain.
2. To investigate tDCS induced functional changes in the brain by using fMRI.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia (ACR-90 criteria, M79.7 ICD10)
* Mean VAS > 4 daily 2 weeks prior to study).

Exclusion Criteria:

* Severe mental disease
* CNS disease
* Mental retardation
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Perceived pain | Change in VAS from baseline up to 49 days.
  Pain (intensity and unpleasentness) measured with Visual Analog Scale. Repported at 3 points daily (0900hrs, 1500hrs, 2100hrs) using Short Message System (SMS) 14 days pre-treatment (baseline), during treatment 5 days, and 30 days post-treatment. Measure effect of active\sham tDCS on pain. 2 levels of group (active tDCS\ sham tDCS, 7 repeated measures: pre-treatment day 1, 2 ,3, 4, 5 - post) SMS messages contain 4 questions, mesauring pain intensity / pain unpleasentness (primary outcome), and stress / activation (secondary outcome).

SECONDARY OUTCOMES:
Cerebral pain processing | Change from baseline to post treatment. 7 days.
  Phillps tesla 1.5 fMRi, pathway pain stimulator (Medoc, Israel) fMRI under pain stimulation for 60 participants. 20 recieve active tDCS, 20 recieve sham-tDCS, 20 age and gender matched (matched to active tDCS group) healthy controls. Baseline scan, post treatment scan.
Rating scales (HADS, SCL90, SF36, FIQ) | Change from baseline to post treatment. 30 days post treatment. Up to 65 days.
  Time from inclusion to treatment start determines 30\14 days. Rating scales on Samsung Galaxy tab 10.1. HADS mesure anxiety and depression, SCL 90 measure symtoms of mental illness, SF36 mesure health related life quality, FIQ mesure symptom severity in fibromyalgia.
Perceived pain, natural history | Baseline compared to post-treatment. Up to 65 days
  Pain (intensity and unpleasentness) measured with Visual Analog Scale. 3 times daily (0900hrs, 1500hrs, 2100hrs). A randomly selected sample of participants have VAS measured with SMS for 30 days pre treatment. Intention is to gather natural history sample to compare with a similarly lengthed post-treatment period.
Perceived stress and activation | Change in VAS from baseline to during treatment and after treatment. Up to 49 days.
  Stress and activation measured with Visual Analog Scale. Repported at 3 points daily (0900hrs, 1500hrs, 2100hrs) using Short Message System (SMS) 14 days pre-treatment (baseline), during treatment 5 days, and 30 days post-treatment. Measure effect of active\sham tDCS on stress and activation. 2 levels of group (active tDCS\ sham tDCS, 7 repeated measures: pre-treatment day 1, 2 ,3, 4, 5 - post) Measured using the same instrumet as the primary outcome.
Perceived stress and activation, natural history | Baseline compared to post-treatment. Up to 65 days
  Stress and activation measured with Visual Analog Scale. 3 times daily (0900hrs, 1500hrs, 2100hrs). A randomly selected sample of participants have VAS measured with SMS for 30 days pre treatment. Intention is to gather natural history sample to compare with a similarly lengthed post-treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Per Aslaksen, ph.d, Study Chair — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Tromsoe, Norway